CLINICAL TRIAL: NCT03363685
Title: An Observational Study of Novel Survival Prediction Algorithm as Clinical Decision Support for Patients With Non-Small-Cell Lung Cancer (NSCLC) Spinal Metastasis
Brief Title: Verification of Novel Survival Prediction Algorithm for Patients With NSCLC Spinal Metastasis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Yuhui Shen, Associate Chief Physician of Orthopaedics, Ruijin Hospital
Other Study IDs: RJ2017NO170
Record Dates: First submitted 2017-11-25; First posted 2017-12-06 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Spinal Metastases; Non-Small-Cell Lung Cancer Metastatic
Keywords: Survival Prediction; Spinal Metastases; Non Small Cell Lung Cancer Metastatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Low risk: For NSCLC spinal metastasis patients with 0-3 of novel survival prediction algorithm.
- Intermediate risk: For NSCLC spinal metastasis patients with 4-6 of novel survival prediction algorithm.
- High risk: For NSCLC spinal metastasis patients with 7-10 of novel survival prediction algorithm.

SUMMARY:
The purpose of this study is to learn whether our own made predictive algorithm can be used as a clinical practical decision support for patients with NSCLC spinal metastasis. The scoring system consists of the use of EGFR-TKI, KPS, Age, SCC, CA125 and smoking history. By predicting survival doctors could determine which patients are suitable for palliative therapy.

DETAILED DESCRIPTION:
Investigators have performed a retrospective study on 176 patients with NSCLC spinal metastasis under the oversight of hospital's ethics committee, and investigators found that the use of EGFR-TKI, KPS, Age, SCC, CA125 and smoking history had significant association with survival. Then investigators built a simple, easy to use scoring system based on the features mentioned above. The score was calculated as 1 (for patients didn't receive EGFR-TKI), +2 (for KPS <50%), +1 (for KPS 50-70%), +1 (Age >60years), 2 (SCC ≥1.5ng/ml), +3 (CA125 ≥35 U/ml), +1 (smoking history 1-10/day), +2 (smoking history >10/day), and 0 otherwise. This algorithm was used to divide the patients into low risk (0-3), intermediate risk (4-6), high risk groups (7-10) to predict survival and determine which patients are suitable for palliative therapy. Now investigators wish to register this study to do a further research, in order to verify the accuracy and sensitivity of this algorithm.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis by biopsy: Non-small-cell lung cancer, including non-squamous carcinoma and squamous cell carcinoma.
* Diagnosis through both nucleotide bone scan and MRI or PET-CT: spinal metastasis.
* Age 18-75 years.
* Have been or is about to be treated according to NCCN panel recommendation.

Exclusion Criteria:

* Diagnosis by biopsy: other tumors.
* Irregular follow-up and lost follow-up
* Withdraw from the study for any reason

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with NSCLC spinal metastasis aged 18-75.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2022-11-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
Survival | Every 6 months from date of diagnosis of NSCLC spinal metastasis until the date of death from any cause, assessed up to 3 years
  Accuracy and sensitivity of novel survival prediction algorithm derived from differences between the predicted and actual survival of NSCLC spinal metastasis patients from 3 different risk groups.

SECONDARY OUTCOMES:
Primary and Metastatic Lesions | Every 6 months from date of diagnosis of NSCLC spinal metastasis until the date of death from any cause, assessed up to 3 years
  Differences in the primary and metastatic lesions after therapy according to NCCN suggestion of NSCLC spinal metastasis patients from 3 different risk groups.
Serum Markers | Every 6 months from date of diagnosis of NSCLC spinal metastasis until the date of death from any cause, assessed up to 3 years
  Differences in the serum markers after therapy according to NCCN suggestion of NSCLC spinal metastasis patients from 3 different risk groups.
Visceral Metastasis | Every 6 months from date of diagnosis of NSCLC spinal metastasis until the date of death from any cause, assessed up to 3 years
  The correlation between visceral metastasis and overall survival (OS) of NSCLC spinal metastasis patients
Visual Analogue Scale (VAS) | Every 6 months from date of diagnosis of NSCLC spinal metastasis until the date of death from any cause, assessed up to 3 years
  Assessment of pain level (1-10, higher value represents more pain)
Ambulatory Status | Every 6 months from date of diagnosis of NSCLC spinal metastasis until the date of death from any cause, assessed up to 3 years
  Assessment of walking ability
EORTC Quality of Life Questionnaire (QLQ) Bone metastasis (BM) 22, | Every 6 months from date of diagnosis of NSCLC spinal metastasis until the date of death from any cause, assessed up to 3 years
  Assessment of quality of life (22-88, higher value represents worse quality of life)
Modified Frankel grade | Every 6 months from date of diagnosis of NSCLC spinal metastasis until the date of death from any cause, assessed up to 3 years
  Assessment of neurological function (A-E, higher value represents better function)
The Spinal Instability Neoplastic Score (SINS) | Every 6 months from date of diagnosis of NSCLC spinal metastasis until the date of death from any cause, assessed up to 3 years
  Assessment of spinal instability (0-18, higher value represents worse instability)

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zang S, He Q, Bao Q, Shen Y, Zhang W. Establishment and validation of a novel survival prediction scoring algorithm for patients with non-small-cell lung cancer spinal metastasis. Int J Clin Oncol. 2019 Sep;24(9):1049-1060. doi: 10.1007/s10147-019-01452-8. Epub 2019 Apr 26. PMID 31028506